CLINICAL TRIAL: NCT02953990
Title: Self-Management of Chronic Depressive Symptoms in Pregnancy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: HM20006941; 1R15HD086835-01A1 (NIH)
Record Dates: First submitted 2016-10-31; First posted 2016-11-03 (Estimated); Results first posted 2024-03-25 (Actual); Last update posted 2024-03-25 (Actual); Status verified 2024-03

CONDITIONS: Depression
Keywords: Pregnancy; Self-Management; Yoga
MeSH Terms: conditions — Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- MOMS Program (Experimental): The MOMS Program involves: (1) mindfulness of symptoms and goal-setting through a nurse-participant partnership, and (2) 12 weeks of weekly community-based group prenatal yoga classes (75 minutes each) and self-directed home activity. Participants will engage in 12 weeks of weekly community-based group prenatal yoga classes (75 minutes each) and self-directed home practice.
  Interventions: Behavioral: MOMS Program

INTERVENTIONS:
Behavioral: MOMS Program

SUMMARY:
This study will provide information about the feasibility, acceptability, and preliminary effects of a biobehavioral self-management approach for perinatal depressive symptoms. This line of research will contribute to the body of knowledge about adjunctive therapies for depressive symptoms in pregnancy, a serious problem which contributes to poor maternal-child outcomes. Ultimately, this will contribute to the development and implementation of theoretically driven depression prevention/ resiliency building interventions and measurement of appropriate biobehavioral outcomes to determine the effectiveness of interventions.

DETAILED DESCRIPTION:
The investigators longitudinal mixed-methods study will use a one-group repeated measures intervention design coupled with qualitative methods to provide a comprehensive view of the feasibility, acceptability, and preliminary effects of the MOMS intervention. Semi-structured interviews, recruitment and retention numbers, and participant logs will be used to evaluate feasibility and acceptability of the intervention (Specific Aim 1). Recently collected archival comparison group data from an existing study will be used to contribute to explorations of preliminary effects of the intervention by comparing longitudinal psychobehavioral data, birth weight data (Specific Aims 2 and 3).

ELIGIBILITY:
Inclusion Criteria:

* ≥ age 18;
* self-report of depressive symptoms prior to pregnancy;
* current depressive symptoms at a moderate-to-severe level, as defined by a score ≥10 on the Patient Health Questionnaire-9;
* able to read, write, and understand English;
* self-identify as black/African American (AA) or White;
* absence of suicidal ideations (measured as low risk on the M.I.N.I. Neuropsychiatric Interview tool);
* absence of pregnancy complications/physical conditions making physical activity (PA) inadvisable;
* has not engaged in a consistent mindfulness-based PA routine during the pregnancy (such as yoga or similar activities more than once per month).

Exclusion Criteria:

* If individual does not meet the inclusion criteria listed above, they are ineligible for the study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2016-09; Primary Completion 2019-02-12 (Actual); Study Completion 2019-02-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Patricia A Kinser, PhD, Principal Investigator — Virginia Commonwealth University
Locations (1):
- Virginia Commonwealth University School of Nursing, Richmond, Virginia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kinser PA, Thacker LR, Rider A, Moyer S, Amstadter AB, Mazzeo SE, Bodnar-Deren S, Starkweather A. Feasibility, Acceptability, and Preliminary Effects of "Mindful Moms": A Mindful Physical Activity Intervention for Pregnant Women with Depression. Nurs Res. 2021 Mar-Apr 01;70(2):95-105. doi: 10.1097/NNR.0000000000000485. PMID 33630532

RESULTS

PARTICIPANT FLOW:
Groups:
- MOMS Program: The MOMS Program involves: (1) mindfulness of symptoms and goal-setting through a nurse-participant partnership, and (2) 12 weeks of weekly community-based group prenatal yoga classes (75 minutes each) and self-directed home activity. Participants will engage in 12 weeks of weekly community-based group prenatal yoga classes (75 minutes each) and self-directed home practice.
  MOMS Program
Period: Overall Study
Arm/Group | MOMS Program
Started | 41
Completed | 27
Not Completed | 14

BASELINE CHARACTERISTICS:
Arm/Group | MOMS Program
Number analyzed (Participants) | 41
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 41
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 29.10 (5.32)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 41
  Male | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 26
  White | 12
  More than one race | 0
  Unknown or Not Reported | 3
Region of Enrollment [Number; unit: participants]
  United States | 41

OUTCOME MEASURES:

1. Primary Outcome: Recruitment Data
Description: # individuals who enrolled in study/ # individuals who expressed interest in the study
Time Frame: baseline
Population: 41 enrolled/ 50 eligible
Measure: Count of Participants; unit: Participants
Arm/Group | MOMS Program
Number analyzed (Participants) | 50
Participants | 41

2. Primary Outcome: Retention Data
Description: # of participants enrolled/ # of participants completing study
Time Frame: 18 weeks post-baseline
Population: 41 enrolled/ 27 completed
Measure: Count of Participants; unit: Participants
Arm/Group | MOMS Program
Number analyzed (Participants) | 41
Participants | 27

3. Primary Outcome: Adherence
Description: Measure of those who attended at least 50% of the yoga sessions (measured analyzing class rosters)
Time Frame: End of 12 week intervention
Measure: Count of Participants; unit: Participants
Arm/Group | MOMS Program
Number analyzed (Participants) | 27
Participants | 26

4. Primary Outcome: Completed Interviews
Description: The number of participants who completed the intervention and completed a postpartum semi-structured interview
Time Frame: End of 6 week postpartum visit
Measure: Count of Participants; unit: Participants
Arm/Group | MOMS Program
Number analyzed (Participants) | 27
Participants | 26

5. Primary Outcome: Edinburgh Postnatal Depression Scale (EPDS)
Description: Pregnancy-specific Depressive Symptoms/Perinatal-specific depressive symptoms were measured by the 10-item Edinburgh Postnatal Depression Scale (EPDS; Cox et al., 1987); scores range from0 to 30, and a score of≥10 is considered indicative of possible depressive symptoms.
Time Frame: baseline and end of 12 week intervention
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | MOMS Program
Number analyzed (Participants) | 27
score on a scale
  Baseline | 15.2 (0.86)
  End of Intervention | 5.05 (0.67)

6. Secondary Outcome: Patient Health Questionnaire-9 (PHQ9)
Description: Depressive Symptoms/ Perceived stress was measured with the 10-item Perceived Stress Scale; scores range from 0 to 40, and higher scores represent higher perceived stress.
Time Frame: baseline and end of 12 week intervention
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | MOMS Program
Number analyzed (Participants) | 27
score on a scale
  Baseline | 13.54 (0.40)
  End of intervention | 5.05 (0.67)

7. Secondary Outcome: State-Trait Anxiety Inventory-State (STAI-S)
Description: State Anxiety/ Anxiety was measured with the State Anxiety Form Y ; scores range from20 to 80, and higher scores indicate higher state anxiety.
Time Frame: baseline and at the end of the 12 week intervention
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | MOMS Program
Number analyzed (Participants) | 27
score on a scale
  Baseline | 50.02 (2.10)
  End of intervention | 36.04 (2.10)

8. Secondary Outcome: Ruminations Response Scale (RRS-10)
Description: Ruminations/ The Ruminative Responses Scale was used to measure ruminations; total scores range from 10 to 40, where higher scores indicate higher rumination.
Time Frame: baseline and at the end of the 12 week intervention
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | MOMS Program
Number analyzed (Participants) | 27
score on a scale
  Baseline | 26.63 (1.08)
  End of intervention | 23.14 (1.29)

9. Secondary Outcome: Self-Efficacy for Physical Activity
Description: Self-Efficacy for Physical Activity: The Physical Activity Self-Efficacy Scale is an eight-question scale that contains items about self-management of physical activities and social support regarding physical activity. A higher score indicates higher self-efficacy. The scores may range form 0-90
Time Frame: Baseline visit to end of 12 week intervention visit
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | MOMS Program
Number analyzed (Participants) | 27
score on a scale
  baseline | 26.04 (7.4)
  end of intervention | 28.6 (7.8)

10. Secondary Outcome: Maternal Fetal Attachment Scale (MFAS)
Description: Maternal-Child Attachment/ Maternal-fetal/ child attachment was measured using the Maternal-Fetal Attachment Scale with wording adapted slightly for the postpartum use; scores range from 24 to 120,with higher scores indicating higher attachment.
Time Frame: baseline and at the end of the 12 week intervention
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | MOMS Program
Number analyzed (Participants) | 27
score on a scale
  Baseline | 54.56 (2.51)
  End of intervention | 43.97 (2.01)

11. Secondary Outcome: Baby's Birth Weight
Description: Baby's birth weight in pounds per mother's report at postpartum visit
Time Frame: postpartum visit
Measure: Mean (Standard Deviation); unit: pounds
Arm/Group | MOMS Program
Number analyzed (Participants) | 21
pounds | 7.57 (1.33)

12. Secondary Outcome: Stress
Description: Perceived Stress Scale (PSS): 10-item scale; scores range from 0 to 40, and higher scores represent higher perceived stress
Time Frame: Change from Baseline visit to end of 12 week intervention visit
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | MOMS Program
Number analyzed (Participants) | 27
score on a scale
  Baseline | 25.27 (0.89)
  End of intervention | 16.72 (1.17)

13. Secondary Outcome: Total # of Minutes in Physical Activity (Including Yoga)
Description: Adherence to physical activity aspect of intervention (including yoga)
Time Frame: End of 12 week intervention
Measure: Mean (Full Range); unit: minutes per week
Arm/Group | MOMS Program
Number analyzed (Participants) | 27
minutes per week | 141 [0 to 1070]

ADVERSE EVENTS:
Time Frame: 18 weeks
Arm/Group | MOMS Program
All-Cause Mortality (participants affected / at risk) | 0/41
Serious Adverse Events (participants affected / at risk) | 0/41
Other Adverse Events (participants affected / at risk) | 0/41

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-04-07): https://cdn.clinicaltrials.gov/large-docs/90/NCT02953990/Prot_SAP_000.pdf